CLINICAL TRIAL: NCT04518995
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of CTP-543 in Adult Patients With Moderate to Severe Alopecia Areata (THRIVE-AA1)
Brief Title: Study to Evaluate the Efficacy and Safety of CTP-543 in Adults With Moderate to Severe Alopecia Areata (THRIVE-AA1)
Acronym: THRIVE-AA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP543.3001; 2020-002704-40 (EudraCT Number)
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Alopecia Areata
Keywords: Alopecia; Hair loss; Hair disease; CTP-543
MeSH Terms: conditions — Alopecia Areata; Alopecia; Hair Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): Participants received CTP-543 matched placebo tablets, orally, twice daily (BID) for up to 24 weeks.
  Interventions: Drug: CTP-543 matching placebo
- CTP-543 8 mg BID (Experimental): Participants received CTP-543 8 mg tablets, orally, BID for up to 24 weeks.
  Interventions: Drug: CTP-543
- CTP-543 12 mg BID (Placebo Comparator): Participants received CTP-543 12 mg tablets, orally, BID for up to 24 weeks.
  Interventions: Drug: CTP-543

INTERVENTIONS:
Drug: CTP-543 matching placebo — Administered as tablets.
  Arms: Placebo
Drug: CTP-543 — Administered as tablets.
  Arms: CTP-543 8 mg BID
Drug: CTP-543 — Administered as tablets.
  Arms: CTP-543 12 mg BID

SUMMARY:
This study evaluates the safety and effectiveness of an investigational study drug (called CTP-543) in adults (18 years and older) who have 50% or greater scalp hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation compatible with alopecia areata with a current episode lasting at least 6 months and not exceeding 10 years at the time of Screening. Total disease duration greater than 10 years is permitted.
* At least 50% scalp hair loss, as defined by a Severity of Alopecia Tool (SALT) score ≥50, at Screening and Baseline.
* Willing to comply with the study visits and requirements of the study protocol.

Exclusion Criteria:

* Treatment with other medications or agents within 1 month of Baseline or during the study that may affect hair regrowth or immune response.
* Active scalp inflammation, psoriasis, or seborrheic dermatitis requiring topical treatment to the scalp, significant trauma to the scalp, or other scalp condition that may interfere with the SALT assessment, or untreated actinic keratosis anywhere on the body at Screening and/or Baseline.
* Treatment with systemic immunosuppressive medications within 3 months of Screening or during the study, or biologics within 6 months of Screening or during the study.
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study drug.
* Clinically significant medical condition, psychiatric disease, or social condition, as determined by the Investigator, that may unfavorably alter the risk-benefit of study participation, adversely affect study compliance, or confound interpretation of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (47):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Kern Research, Inc., Bakersfield, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - UC Irvine Dermatology Clinical Research Center, Irvine, California
  - Quest Dermatology Research, Northridge, California
  - Kaiser Permanente, Oakland, California
  - Kaiser Permanente South Sacramento, Sacramento, California
  - Kaiser Permanente, San Francisco, California
  - Colorado Center for Dermatology and Skin Surgery, Centennial, Colorado
  - Colorado Medical Research Center, Denver, Colorado
  - Yale University, Church Street Research Unit, New Haven, Connecticut
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Forward Clinical Trials Inc., Tampa, Florida
  - Denova Research, Chicago, Illinois
  - Northwestern Memorial Hospital, Department of Dermatology, Chicago, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DS Research, New Albany, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - DS Research, Louisville, Kentucky
  - Qualmedica Research LLC, Owensboro, Kentucky
  - Massachusetts General Hospital - Clinic, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clarkston Skin Research, Clarkston, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - University of Minnesota Department of Dermatology, Minneapolis, Minnesota
  - Skin Laser and Surgery Specialists of NJ, Hackensack, New Jersey
  - Sadick Research Group, New York, New York
  - Darst Dermatology, Charlotte, North Carolina
  - Dermatology Specialists of Charlotte, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Department of Dermatology, Winston-Salem, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Northwest Dermatology Institute, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Dermatology Associates Of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - PEAK Research, Upper Saint Clair, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Palmetto Clinical Trial Services, Fountain Inn, South Carolina
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Austin Institute for Clinical Research, Inc., Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - West End Dermatology Associates, Richmond, Virginia
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
- Canada (14):
  - Dermatology Research Institute, Calgary, Alberta
  - Kirk Barber Research, Calgary, Alberta
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Dr Wei Jing Loo Medicine Professional Corporation, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - JRB Research Inc., Ottawa, Ontario
  - Research Toronto, Toronto, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - Innovaderm Research Inc. - Clinic, Montreal, Quebec
- France (5):
  - Hôpital Saint-André - Chu de Bordeaux, Bordeaux, Nouvelle-Aquitaine
  - Hôpital Saint-Louis - Gh de La Rochelle, La Rochelle, Nouvelle-Aquitaine
  - Hôpital Hotel Dieu - Chu de Nantes, Nantes, Pays de la Loire Region
  - Hôpital La Timone-Dermatologie, Marseille
  - Hôpital Saint Louis, Centre de Santé Sabouraud, Paris
- Poland (4):
  - Vita Longa Sp.Zo.O, Katowice
  - SGD S.C., Krakow
  - My Clinic, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
- Spain (2):
  - Hospital Clínico Y Provincial de Barcelona, Barcelona
  - H. U. Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in Canada, France, Poland, Spain and the United States from 23 November 2020 to 19 April 2022.
Pre-assignment Details: 946 participants were screened, out of which 706 participants who experienced moderate to severe hair loss due to alopecia areata were enrolled to receive CTP-543 or placebo.
Period: Overall Study
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Started | 140 | 351 | 215
Efficacy Population (Efficacy population included all participants who were randomized in the study and dispensed study drug during the treatment period.) | 140 | 351 | 215
Safety Population (Safety population included all participants who received study drug during the treatment period.) | 140 | 350 | 215
Completed | 129 | 318 | 199
Not Completed | 11 | 33 | 16
Not completed — Treatment Emergent or Worsening Adverse Event | 2 | 8 | 4
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Non-compliance With Study Drug | 0 | 3 | 2
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 1
Not completed — Reason not Specified | 4 | 11 | 2
Not completed — Lost to Follow-up | 1 | 10 | 6

BASELINE CHARACTERISTICS:
Population: All randomized participants included all participants who were randomized in the study.
Groups:
- Placebo: Participants received CTP-543 matched placebo tablets, orally, BID for up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID | Total
Number analyzed (Participants) | 140 | 351 | 215 | 706
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (13.81) | 38.9 (13.32) | 38.2 (12.80) | 38.6 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 217 | 131 | 437
  Male | 51 | 134 | 84 | 269
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 30 | 13 | 54
  Not Hispanic or Latino | 119 | 292 | 188 | 599
  Unknown or Not Reported | 10 | 29 | 14 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 2 | 1 | 3
  Race: Asian | 10 | 22 | 21 | 53
  Race: Black or African American | 16 | 40 | 27 | 83
  Race: Native Hawaiian or other Pacific Islander | 1 | 3 | 1 | 5
  Race: White | 98 | 241 | 145 | 484
  Race: Other | 5 | 17 | 6 | 28
  Race: Not reported | 10 | 26 | 14 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Absolute Severity of Alopecia Tool (SALT) Score of ≤20 at Week 24
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss).
Time Frame: Week 24
Population: Efficacy population included all participants who were randomized in the study and dispensed study drug during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 140 | 351 | 215
percentage of participants | 0.8 | 29.6 | 41.5
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Test type: Superiority; p < 0.0001, Mantel Haenszel — P-value was calculated by Mantel-Haenszel estimate stratified by baseline scalp hair loss (partial vs complete/near-complete) for each treatment group compared to placebo; Risk Difference (RD) = 0.28, 95% CI 2-sided [0.23 to 0.33], Standard Error of Mean 0.026
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.39, 95% CI 2-sided [0.32 to 0.46], Standard Error of Mean 0.034

2. Secondary Outcome: Percentage of Responders on the Hair Satisfaction Patient Reported Outcome (SPRO) Scale at Weeks 12, 16, 20, and 24
Description: SPRO is a questionnaire answered by the participant and designed to measure how satisfied alopecia areata participants are with their hair at the time of the assessment. The responses range from 1 to 5: 1= very satisfied, 2= satisfied, 3= neither satisfied nor dissatisfied, 4= dissatisfied, and 5= very dissatisfied. Responders were defined as participants with responses of "satisfied" or "very satisfied".
Time Frame: Weeks 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 140 | 351 | 215
percentage of responders
  Week 12 | 11.9 | 35.3 | 46.4
  Week 16 | 8.3 | 38.2 | 51.5
  Week 20 | 6.1 | 37.4 | 54.0
  Week 24 | 4.7 | 42.1 | 53.0
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.25, 95% CI 2-sided [0.17 to 0.32], Standard Error of Mean 0.038
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.35, 95% CI 2-sided [0.26 to 0.43], Standard Error of Mean 0.044
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.31, 95% CI 2-sided [0.24 to 0.38], Standard Error of Mean 0.035
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.43, 95% CI 2-sided [0.35 to 0.51], Standard Error of Mean 0.041
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.32, 95% CI 2-sided [0.26 to 0.39], Standard Error of Mean 0.033
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.47, 95% CI 2-sided [0.39 to 0.55], Standard Error of Mean 0.040
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.38, 95% CI 2-sided [0.31 to 0.44], Standard Error of Mean 0.033
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.47, 95% CI 2-sided [0.39 to 0.55], Standard Error of Mean 0.039

3. Secondary Outcome: Percentage of Participants Achieving an Absolute SALT Score of ≤20 at Weeks 4, 8, 12, 16, and 20
Description: as for outcome 1
Time Frame: Weeks 4, 8, 12, 16, and 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 140 | 351 | 215
percentage of participants
  Week 4 | 0 | 0.9 | 0
  Week 8 | 0 | 3.3 | 6.1
  Week 12 | 0.7 | 10.4 | 18.2
  Week 16 | 2.3 | 16.5 | 29.6
  Week 20 | 0.8 | 24.1 | 37.0
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 4; Test type: Superiority; p = 0.0816, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.01, 95% CI 2-sided [-0.00 to 0.02], Standard Error of Mean 0.005
Statistical Analysis 2: Comparison: Placebo vs CTP-543 8 mg BID; Week 8; Test type: Superiority; p = 0.0005, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.03, 95% CI 2-sided [0.01 to 0.05], Standard Error of Mean 0.010
Statistical Analysis 3: Comparison: Placebo vs CTP-543 12 mg BID; Week 8; Test type: Superiority; p = 0.0002, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.06, 95% CI 2-sided [0.03 to 0.09], Standard Error of Mean 0.016
Statistical Analysis 4: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.10, 95% CI 2-sided [0.06 to 0.14], Standard Error of Mean 0.018
Statistical Analysis 5: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.17, 95% CI 2-sided [0.12 to 0.22], Standard Error of Mean 0.027
Statistical Analysis 6: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.14, 95% CI 2-sided [0.10 to 0.19], Standard Error of Mean 0.024
Statistical Analysis 7: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.27, 95% CI 2-sided [0.20 to 0.33], Standard Error of Mean 0.033
Statistical Analysis 8: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.23, 95% CI 2-sided [0.19 to 0.28], Standard Error of Mean 0.024
Statistical Analysis 9: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.35, 95% CI 2-sided [0.28 to 0.41], Standard Error of Mean 0.034

4. Secondary Outcome: Relative Change in SALT Scores From Baseline at Weeks 4, 8, 12, 16, 20, and 24
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss). Relative change (percent change) to baseline is calculated as: 100 x ([post-baseline SALT score - baseline SALT score]/baseline SALT score).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Efficacy population included all participants who were randomized in the study and dispensed study drug during the treatment period. Overall number of participants analyzed indicates the number of participants with data available for analysis of this outcome measure. Number of participants analyzed indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 139 | 345 | 212
percent change
  Relative Change From Baseline at Week 4: number analyzed (Participants) | 139 | 345 | 211
  Relative Change From Baseline at Week 4 | -0.2 (5.59) | -2.6 (12.79) | -4.0 (12.03)
  Relative Change From Baseline at Week 8: number analyzed (Participants) | 138 | 336 | 212
  Relative Change From Baseline at Week 8 | -2.3 (11.41) | -10.9 (21.00) | 17.5 (27.16)
  Relative Change From Baseline at Week 12: number analyzed (Participants) | 136 | 328 | 209
  Relative Change From Baseline at Week 12 | -0.6 (16.63) | -22.2 (29.45) | -31.1 (35.53)
  Relative Change From Baseline at Week 16: number analyzed (Participants) | 131 | 322 | 203
  Relative Change From Baseline at Week 16 | -1.8 (21.06) | -30.3 (34.20) | -41.2 (38.95)
  Relative Change From Baseline at Week 20: number analyzed (Participants) | 131 | 316 | 200
  Relative Change From Baseline at Week 20 | -1.3 (22.14) | -36.0 (37.82) | -46.8 (41.32)
  Relative Change From Baseline at Week 24: number analyzed (Participants) | 128 | 318 | 200
  Relative Change From Baseline at Week 24 | -1.5 (23.30) | -41.2 (39.37) | -50.4 (41.52)
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 4; Test type: Superiority; p = 0.0564, MMRM — P-value was calculated by mixed model repeated measures (MMRM) analysis with effects for treatment, visit, treatment-by-visit interaction, and baseline value; Least Square (LS) Mean Difference = -2.2, 95% CI 2-sided [-4.4 to 0.1], Standard Error of Mean 1.13
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 4; Test type: Superiority; p = 0.0054, MMRM — P-value was calculated by MMRM analysis with effects for treatment, visit, treatment-by-visit interaction, and baseline value; LS Mean Difference = -3.4, 95% CI 2-sided [-5.9 to -1.0], Standard Error of Mean 1.23
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 8; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -8.5, 95% CI 2-sided [-12.7 to -4.3], Standard Error of Mean 2.16
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 8; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -14.9, 95% CI 2-sided [-19.5 to -10.3], Standard Error of Mean 2.34
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -21.7, 95% CI 2-sided [-27.5 to -16.0], Standard Error of Mean 2.94
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -30.0, 95% CI 2-sided [-36.3 to -23.8], Standard Error of Mean 3.19
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -28.4, 95% CI 2-sided [-35.1 to -21.8], Standard Error of Mean 3.38
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -38.5, 95% CI 2-sided [-45.7 to -31.3], Standard Error of Mean 3.66
Statistical Analysis 9: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -34.9, 95% CI 2-sided [-42.1 to -27.7], Standard Error of Mean 3.66
Statistical Analysis 10: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -44.6, 95% CI 2-sided [-52.3 to -36.8], Standard Error of Mean 3.96
Statistical Analysis 11: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -39.3, 95% CI 2-sided [-46.7 to -31.8], Standard Error of Mean 3.79
Statistical Analysis 12: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -47.0, 95% CI 2-sided [-55.1 to -39.0], Standard Error of Mean 4.10

5. Secondary Outcome: Percentage of Responders Assessed Using the Clinician Global Impression of Improvement (CGI-I) at Weeks 12, 16, 20, and 24
Description: The CGI-I is a questionnaire that asks the clinician to evaluate the improvement or worsening of the participant's alopecia areata as compared to the start of the study on a 7-point scale. Responses range from 1 (very much worse) to 7 (very much improved). Responders were defined as participants with responses of 6 (much improved) or 7 (very much improved).
Time Frame: Weeks 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 140 | 351 | 215
percentage of responders
  Week 12 | 3.7 | 36.3 | 43.5
  Week 16 | 7.7 | 44.2 | 54.7
  Week 20 | 8.4 | 49.1 | 57.1
  Week 24 | 9.4 | 53.8 | 59.8
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated by cochran mantel haenszel (CMH) test stratified by baseline scalp hair loss (partial vs complete/near-complete) for responders in each treatment group compared to placebo
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated by CMH test stratified by baseline scalp hair loss (partial vs complete/near-complete) for responders in each treatment group compared to placebo
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]

6. Secondary Outcome: Percentage of Responders Assessed Using the Patient Global Impression of Improvement (PGI-I) at Weeks 12, 16, 20, and 24
Description: The PGI-I is a self-administered questionnaire that asks the participant to evaluate the improvement or worsening of their alopecia areata as compared to the start of the study on a 7-point scale. Responses range from 1 (very much worse) to 7 (very much improved). Responders were defined as participants with responses of 6 (much improved) or 7 (very much improved).
Time Frame: Weeks 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 140 | 351 | 215
percentage of responders
  Week 12 | 6.7 | 38.9 | 49.8
  Week 16 | 9.0 | 49.1 | 58.3
  Week 20 | 10.0 | 50.6 | 60.0
  Week 24 | 10.2 | 56.6 | 65.5
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]

7. Secondary Outcome: Change in the Clinician Global Impression of Severity (CGI-S) Scores From Baseline at Weeks 12, 16, 20, and 24
Description: The CGI-S is a questionnaire that asks the clinician to evaluate the symptom severity of the participant's alopecia areata at the time of assessment. The symptom severity was rated on a scale ranging from 1 to 7, where 1=normal, no hair loss; 2=borderline hair loss; 3=mild hair loss; 4=moderate hair loss; 5=marked hair loss; 6=severe hair loss; 7=among the most extreme hair loss. Higher scores indicate more hair loss. A negative change from baseline indicates less hair loss.
Time Frame: Baseline, Weeks 12, 16, 20, and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 136 | 328 | 209
score on a scale
  Baseline | 6.5 (0.74) | 6.4 (0.86) | 6.4 (0.76)
  Change From Baseline at Week 12: number analyzed (Participants) | 136 | 327 | 209
  Change From Baseline at Week 12 | -0.1 (0.74) | -1.0 (1.38) | -1.4 (1.53)
  Change From Baseline at Week 16: number analyzed (Participants) | 131 | 321 | 203
  Change From Baseline at Week 16 | -0.2 (0.99) | -1.3 (1.55) | -1.9 (1.77)
  Change From Baseline at Week 20: number analyzed (Participants) | 131 | 314 | 200
  Change From Baseline at Week 20 | -0.1 (0.83) | -1.6 (1.77) | -2.2 (1.92)
  Change From Baseline at Week 24: number analyzed (Participants) | 127 | 317 | 200
  Change From Baseline at Week 24 | -0.2 (0.90) | -1.9 (1.89) | -2.4 (2.03)
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — P-value was calculated by MMRM analysis with effects for treatment, visit, treatment-by-visit interaction, baseline value, and baseline SALT score; LS Mean Difference = -0.9, 95% CI 2-sided [-1.2 to -0.7], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-1.5 to -0.9], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-1.4 to -0.9], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.6, 95% CI 2-sided [-1.9 to -1.3], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-1.8 to -1.2], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-2.3 to -1.6], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.7, 95% CI 2-sided [-2.0 to -1.3], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-2.5 to -1.7], Standard Error of Mean 0.19

8. Secondary Outcome: Change in the Patient Global Impression of Severity (PGI-S) Scores From Baseline at Weeks 12, 16, 20, and 24
Description: The PGI-S is a self-administered questionnaire that asks the participant to evaluate the symptom severity of their alopecia areata at the time of assessment. Symptom severity was rated on a scale ranging from 1 to 7, where 1=normal, no hair loss; 2=borderline hair loss; 3=mild hair loss; 4=moderate hair loss; 5=marked hair loss; 6=severe hair loss; 7=among the most extreme hair loss. Higher scores indicate more hair loss. A negative change from baseline indicates less hair loss.
Time Frame: Baseline, Weeks 12, 16, 20, and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 137 | 329 | 209
score on a scale
  Baseline | 6.5 (0.76) | 6.5 (0.80) | 6.4 (0.86)
  Change From Baseline at Week 12: number analyzed (Participants) | 135 | 329 | 209
  Change From Baseline at Week 12 | -0.4 (1.08) | -1.1 (1.64) | -1.4 (1.79)
  Change From Baseline at Week 16: number analyzed (Participants) | 133 | 322 | 204
  Change From Baseline at Week 16 | -0.2 (0.78) | -1.5 (1.83) | -2.0 (1.95)
  Change From Baseline at Week 20: number analyzed (Participants) | 130 | 318 | 200
  Change From Baseline at Week 20 | -0.3 (1.01) | -1.8 (2.01) | -2.2 (2.07)
  Change From Baseline at Week 24: number analyzed (Participants) | 128 | 318 | 200
  Change From Baseline at Week 24 | -0.1 (0.74) | -1.9 (2.05) | -2.4 (2.14)
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — P-value was calculated by MMRM with effects for treatment, visit, treatment-by-visit interaction, baseline value, and baseline SALT score; LS Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.3], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-1.3 to -0.6], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-1.6 to -0.9], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.7, 95% CI 2-sided [-2.1 to -1.4], Standard Error of Mean 0.18
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-1.7 to -1.0], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-2.3 to -1.5], Standard Error of Mean 0.20
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.7, 95% CI 2-sided [-2.0 to -1.3], Standard Error of Mean 0.19
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -2.2, 95% CI 2-sided [-2.6 to -1.8], Standard Error of Mean 0.20

9. Secondary Outcome: Percentage of Participants Achieving at Least a 75% and 90% Relative Reduction in SALT Score From Baseline at Weeks 12 and 24
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss). Percentage of participants achieving at least a 75% and 90% relative reduction in SALT score from baseline at Weeks 12 and 24 are reported.
Time Frame: Baseline, Weeks 12, and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 140 | 351 | 215
percentage of participants
  75% Relative Reduction: Week 12 | 0 | 8.8 | 17.7
  75% Relative Reduction: Week 24 | 0 | 28.6 | 40.0
  90% Relative Reduction: Week 12 | 0 | 3.4 | 10.0
  90% Relative Reduction: Week 24 | 0 | 19.2 | 32.0
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; 75% Relative Reduction: Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.09, 95% CI 2-sided [0.06 to 0.12], Standard Error of Mean 0.016
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; 75% Relative Reduction: Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.17, 95% CI 2-sided [0.12 to 0.22], Standard Error of Mean 0.026
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; 75% Relative Reduction: Week 24; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.28, 95% CI 2-sided [0.23 to 0.33], Standard Error of Mean 0.025
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; 75% Relative Reduction: Week 24; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.38, 95% CI 2-sided [0.32 to 0.45], Standard Error of Mean 0.033
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; 90% Relative Reduction: Week 12; Test type: Superiority; p = 0.0006, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.04, 95% CI 2-sided [0.02 to 0.06], Standard Error of Mean 0.010
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; 90% Relative Reduction: Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.10, 95% CI 2-sided [0.06 to 0.14], Standard Error of Mean 0.020
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; 90% Relative Reduction: Week 24; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.19, 95% CI 2-sided [0.15 to 0.23], Standard Error of Mean 0.022
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; 90% Relative Reduction: Week 24; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.30, 95% CI 2-sided [0.24 to 0.37], Standard Error of Mean 0.032

10. Secondary Outcome: Change in the Brigham Eyebrow Tool for Alopecia (BETA) Scores From Baseline at Weeks 12 and 24
Description: BETA is a clinician-rated scale that assesses the total eyebrow hair present. The BETA score is calculated based on hair density and surface area of each individual eyebrow of the participant, ranging from 0 to 3, where 0 = no eyebrow, 1 = minimal eyebrow, 2 = moderate eyebrow, 3 = normal eyebrow. The BETA score is the sum of the right and left eyebrow scores, ranging from 0 to 6. Higher scores indicate less hair loss of eyebrows. A positive change from baseline indicates less hair loss of eyebrows.
Time Frame: Baseline, Weeks 12, and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 83 | 204 | 132
score on a scale
  Baseline | 1.7 (2.05) | 1.2 (1.77) | 1.4 (1.91)
  Change From Baseline at Week 12: number analyzed (Participants) | 76 | 187 | 123
  Change From Baseline at Week 12 | -0.2 (1.38) | 0.8 (1.70) | 1.1 (2.05)
  Change From Baseline at Week 24: number analyzed (Participants) | 72 | 192 | 118
  Change From Baseline at Week 24 | -0.2 (1.68) | 1.6 (1.96) | 1.8 (2.17)
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p = 0.0010, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = 0.7, 95% CI 2-sided [0.3 to 1.2], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = 1.1, 95% CI 2-sided [0.6 to 1.6], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = 1.7, 95% CI 2-sided [1.2 to 2.2], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = 1.9, 95% CI 2-sided [1.4 to 2.4], Standard Error of Mean 0.26

11. Secondary Outcome: Change in the Brigham Eyelash Tool for Alopecia (BELA) Scores From Baseline at Weeks 12 and 24
Description: BELA is a clinician-rated scale that assesses the total eyelash hair present. The BELA is calculated based on distribution and grade values, ranging from 0 (no eyelashes) to 3 (full eyelashes). The BELA score is the sum of the individual scores for the left and right eyes, ranging from 0 to 6. Higher scores indicate less hair loss of eyelashes. A positive change from baseline indicates less hair loss of eyelashes.
Time Frame: Baseline, Weeks 12, and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 86 | 219 | 150
score on a scale
  Baseline | 1.5 (2.12) | 1.4 (2.10) | 1.7 (2.12)
  Change From Baseline at Week 12: number analyzed (Participants) | 84 | 215 | 145
  Change From Baseline at Week 12 | -0.1 (1.18) | 0.9 (1.50) | 1.3 (2.08)
  Change From Baseline at Week 24: number analyzed (Participants) | 78 | 209 | 138
  Change From Baseline at Week 24 | 0.3 (1.30) | 1.7 (1.99) | 2.0 (2.28)
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = 0.9, 95% CI 2-sided [0.5 to 1.3], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = 1.4, 95% CI 2-sided [1.0 to 1.8], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = 1.5, 95% CI 2-sided [1.0 to 2.0], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = 1.9, 95% CI 2-sided [1.4 to 2.4], Standard Error of Mean 0.26

12. Secondary Outcome: Change in the SPRO Scale From Baseline at Weeks 12, 16, 20, and 24
Description: SPRO is a questionnaire answered by the participant and designed to measure how satisfied alopecia areata participants are with their hair at the time of the assessment. The responses range from 1 to 5: 1= very satisfied, 2= satisfied, 3= neither satisfied nor dissatisfied, 4= dissatisfied, and 5= very dissatisfied. Higher scores indicate the greater hair dissatisfaction. A negative change from baseline indicate the greater hair satisfaction.
Time Frame: Baseline, Weeks 12, 16, 20, and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 137 | 329 | 209
score on a scale
  Baseline | 4.5 (0.86) | 4.5 (0.89) | 4.5 (0.85)
  Change From Baseline at Week 12: number analyzed (Participants) | 135 | 329 | 209
  Change From Baseline at Week 12 | -0.6 (1.15) | -1.3 (1.42) | -1.7 (1.36)
  Change From Baseline at Week 16: number analyzed (Participants) | 133 | 322 | 204
  Change From Baseline at Week 16 | -0.4 (1.18) | -1.4 (1.44) | -1.8 (1.43)
  Change From Baseline at Week 20: number analyzed (Participants) | 131 | 318 | 200
  Change From Baseline at Week 20 | -0.4 (1.14) | -1.4 (1.52) | -1.8 (1.52)
  Change From Baseline at Week 24: number analyzed (Participants) | 128 | 318 | 200
  Change From Baseline at Week 24 | -0.3 (1.09) | -1.5 (1.54) | -1.9 (1.64)
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.0 to -0.5], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -1.1, 95% CI 2-sided [-1.3 to -0.8], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -1.0, 95% CI 2-sided [-1.2 to -0.8], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -1.4, 95% CI 2-sided [-1.6 to -1.1], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -1.1, 95% CI 2-sided [-1.3 to -0.8], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -1.5, 95% CI 2-sided [-1.7 to -1.2], Standard Error of Mean 0.14
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -1.2, 95% CI 2-sided [-1.5 to -1.0], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 2]; LS Mean Difference = -1.6, 95% CI 2-sided [-1.8 to -1.3], Standard Error of Mean 0.14

13. Secondary Outcome: Percentage of Participants Achieving a ≥2-point Change From Baseline in the SPRO Scale at Weeks 12, 16, 20, and 24
Description: SPRO is a questionnaire answered by the participant and designed to measure how satisfied alopecia areata participants are with their hair at the time of the assessment. The responses range from 1 to 5: 1= very satisfied, 2= satisfied, 3= neither satisfied nor dissatisfied, 4= dissatisfied, and 5= very dissatisfied.
Time Frame: Weeks 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 140 | 351 | 215
percentage of participants
  Week 12 | 20.7 | 44.7 | 53.1
  Week 16 | 14.3 | 48.1 | 53.9
  Week 20 | 13.7 | 47.5 | 57.5
  Week 24 | 12.5 | 49.1 | 58.0
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — P-value was calculated by the Mantel-Haenszel estimate stratified by baseline scalp hair loss (partial vs complete/near-complete) for each treatment group compared to placebo; Risk Difference (RD) = 0.25, 95% CI 2-sided [0.17 to 0.34], Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Week 12; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.32, 95% CI 2-sided [0.23 to 0.42], Standard Error of Mean 0.049
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Week 16; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.35, 95% CI 2-sided [0.27 to 0.42], Standard Error of Mean 0.040
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Week 16; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.39, 95% CI 2-sided [0.30 to 0.48], Standard Error of Mean 0.045
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Week 20; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.34, 95% CI 2-sided [0.26 to 0.42], Standard Error of Mean 0.040
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Week 20; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.42, 95% CI 2-sided [0.34 to 0.51], Standard Error of Mean 0.045
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Week 24; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.37, 95% CI 2-sided [0.29 to 0.44], Standard Error of Mean 0.039
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Week 24; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.44, 95% CI 2-sided [0.35 to 0.53], Standard Error of Mean 0.045

14. Secondary Outcome: Change in the Individual Items of the Hair Quality Patient Reported Outcome (QPRO) Scale From Baseline at Weeks 12, 16, 20, and 24
Description: The QPRO questionnaire provides additional details on key attributes of hair and helps provide context to the SPRO response. The individual items of QPRO are: Satisfied thickness hair coverage; Satisfied evenness hair coverage; How satisfied with your eyebrows; How satisfied with your eyelashes, scored on a scale ranging from 1 to 5 where 1=very satisfied, 2=satisfied, 3=neither satisfied nor dissatisfied, 4=dissatisfied, 5=very dissatisfied. Higher scores indicate the greater dissatisfaction on hair quality. A negative change from baseline indicate the greater satisfaction on hair quality.
Time Frame: Baseline, Weeks 12, 16, 20, and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 137 | 329 | 209
score on a scale
  Satisfied Thickness Hair Coverage: Baseline | 4.5 (0.79) | 4.6 (0.79) | 4.5 (0.76)
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 12: number analyzed (Participants) | 135 | 329 | 209
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 12 | -0.4 (0.98) | -1.1 (1.23) | -1.3 (1.17)
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 16: number analyzed (Participants) | 133 | 322 | 204
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 16 | -0.3 (1.03) | -1.2 (1.28) | -1.5 (1.33)
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 20: number analyzed (Participants) | 131 | 318 | 200
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 20 | -0.3 (0.98) | -1.3 (1.35) | -1.6 (1.36)
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 24: number analyzed (Participants) | 128 | 318 | 200
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 24 | -0.2 (1.00) | -1.4 (1.43) | -1.7 (1.45)
  Satisfied Evenness Hair Coverage: Baseline | 4.6 (0.67) | 4.6 (0.76) | 4.6 (0.68)
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 12: number analyzed (Participants) | 135 | 329 | 209
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 12 | -0.4 (0.83) | -1.0 (1.19) | -1.3 (1.16)
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 16: number analyzed (Participants) | 133 | 322 | 204
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 16 | -0.3 (0.84) | -1.1 (1.31) | -1.4 (1.34)
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 20: number analyzed (Participants) | 131 | 318 | 200
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 20 | -0.3 (0.90) | -1.2 (1.36) | -1.5 (1.40)
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 24: number analyzed (Participants) | 128 | 318 | 200
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 24 | -0.2 (0.84) | -1.2 (1.41) | -1.6 (1.52)
  How Satisfied With Your Eyebrows: Baseline | 3.8 (1.39) | 4.0 (1.28) | 3.9 (1.35)
  How Satisfied With Your Eyebrows: Change From Baseline at Week 12: number analyzed (Participants) | 135 | 329 | 209
  How Satisfied With Your Eyebrows: Change From Baseline at Week 12 | -0.2 (0.88) | -1.0 (1.20) | -1.1 (1.34)
  How Satisfied With Your Eyebrows: Change From Baseline at Week 16: number analyzed (Participants) | 133 | 322 | 204
  How Satisfied With Your Eyebrows: Change From Baseline at Week 16 | -0.1 (0.90) | -1.1 (1.24) | -1.3 (1.27)
  How Satisfied With Your Eyebrows: Change From Baseline at Week 20: number analyzed (Participants) | 131 | 318 | 200
  How Satisfied With Your Eyebrows: Change From Baseline at Week 20 | -0.2 (0.88) | -1.2 (1.25) | -1.4 (1.32)
  How Satisfied With Your Eyebrows: Change From Baseline at Week 24: number analyzed (Participants) | 128 | 318 | 200
  How Satisfied With Your Eyebrows: Change From Baseline at Week 24 | -0.2 (0.87) | -1.2 (1.26) | -1.4 (1.36)
  How Satisfied With Your Eyelashes: Baseline | 3.7 (1.44) | 3.9 (1.37) | 3.7 (1.44)
  How Satisfied With Your Eyelashes: Change From Baseline at Week 12: number analyzed (Participants) | 135 | 329 | 209
  How Satisfied With Your Eyelashes: Change From Baseline at Week 12 | -0.3 (0.79) | -0.9 (1.21) | -0.9 (1.24)
  How Satisfied With Your Eyelashes: Change From Baseline at Week 16: number analyzed (Participants) | 133 | 322 | 204
  How Satisfied With Your Eyelashes: Change From Baseline at Week 16 | -0.2 (0.97) | -1.0 (1.24) | -1.2 (1.30)
  How Satisfied With Your Eyelashes: Change From Baseline at Week 20: number analyzed (Participants) | 131 | 318 | 200
  How Satisfied With Your Eyelashes: Change From Baseline at Week 20 | -0.3 (0.99) | -1.1 (1.30) | -1.1 (1.33)
  How Satisfied With Your Eyelashes: Change From Baseline at Week 24: number analyzed (Participants) | 128 | 318 | 200
  How Satisfied With Your Eyelashes: Change From Baseline at Week 24 | -0.2 (0.95) | -1.1 (1.37) | -1.2 (1.37)
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Satisfied Thickness Hair Coverage: Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.5], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Satisfied Thickness Hair Coverage: Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.2 to -0.7], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Satisfied Thickness Hair Coverage: Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.6], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Satisfied Thickness Hair Coverage: Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-1.4 to -1.0], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Placebo vs CTP-543 8 mg BID; Satisfied Thickness Hair Coverage: Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-1.2 to -0.8], Standard Error of Mean 0.12
Statistical Analysis 6: Comparison: Placebo vs CTP-543 12 mg BID; Satisfied Thickness Hair Coverage: Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-1.6 to -1.1], Standard Error of Mean 0.13
Statistical Analysis 7: Comparison: Placebo vs CTP-543 8 mg BID; Satisfied Thickness Hair Coverage: Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-1.3 to -0.8], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Placebo vs CTP-543 12 mg BID; Satisfied Thickness Hair Coverage: Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-1.7 to -1.2], Standard Error of Mean 0.14
Statistical Analysis 9: Comparison: Placebo vs CTP-543 8 mg BID; Satisfied Evenness Hair Coverage: Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-0.8 to -0.4], Standard Error of Mean 0.10
Statistical Analysis 10: Comparison: Placebo vs CTP-543 12 mg BID; Satisfied Evenness Hair Coverage: Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.7], Standard Error of Mean 0.11
Statistical Analysis 11: Comparison: Placebo vs CTP-543 8 mg BID; Satisfied Evenness Hair Coverage: Week 16; Test type: Superiority; p < 0.0001, MMRM — P-value was calculated by MMRM mixed model repeated measures analysis with effects for treatment, visit, treatment-by-visit interaction, baseline value, and baseline SALT score; LS Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.5], Standard Error of Mean 0.11
Statistical Analysis 12: Comparison: Placebo vs CTP-543 12 mg BID; Satisfied Evenness Hair Coverage: Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 14, analysis 11]; LS Mean Difference = -1.1, 95% CI 2-sided [-1.3 to -0.8], Standard Error of Mean 0.12
Statistical Analysis 13: Comparison: Placebo vs CTP-543 8 mg BID; Satisfied Evenness Hair Coverage: Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 14, analysis 11]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.7], Standard Error of Mean 0.12
Statistical Analysis 14: Comparison: Placebo vs CTP-543 12 mg BID; Satisfied Evenness Hair Coverage: Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 14, analysis 11]; LS Mean Difference = -1.2, 95% CI 2-sided [-1.5 to -1.0], Standard Error of Mean 0.13
Statistical Analysis 15: Comparison: Placebo vs CTP-543 8 mg BID; Satisfied Evenness Hair Coverage: Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 14, analysis 11]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.2 to -0.7], Standard Error of Mean 0.12
Statistical Analysis 16: Comparison: Placebo vs CTP-543 12 mg BID; Satisfied Evenness Hair Coverage: Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 14, analysis 11]; LS Mean Difference = -1.3, 95% CI 2-sided [-1.5 to -1.0], Standard Error of Mean 0.13
Statistical Analysis 17: Comparison: Placebo vs CTP-543 8 mg BID; How Satisfied With Your Eyebrows: Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.5], Standard Error of Mean 0.11
Statistical Analysis 18: Comparison: Placebo vs CTP-543 12 mg BID; How Satisfied With Your Eyebrows: Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-1.1 to -0.6], Standard Error of Mean 0.12
Statistical Analysis 19: Comparison: Placebo vs CTP-543 8 mg BID; How Satisfied With Your Eyebrows: Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.7], Standard Error of Mean 0.11
Statistical Analysis 20: Comparison: Placebo vs CTP-543 12 mg BID; How Satisfied With Your Eyebrows: Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-1.4 to -0.9], Standard Error of Mean 0.12
Statistical Analysis 21: Comparison: Placebo vs CTP-543 8 mg BID; How Satisfied With Your Eyebrows: Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.7], Standard Error of Mean 0.11
Statistical Analysis 22: Comparison: Placebo vs CTP-543 12 mg BID; How Satisfied With Your Eyebrows: Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-1.3 to -0.9], Standard Error of Mean 0.12
Statistical Analysis 23: Comparison: Placebo vs CTP-543 8 mg BID; How Satisfied With Your Eyebrows: Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-1.2 to -0.8], Standard Error of Mean 0.11
Statistical Analysis 24: Comparison: Placebo vs CTP-543 12 mg BID; How Satisfied With Your Eyebrows: Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-1.4 to -0.9], Standard Error of Mean 0.12
Statistical Analysis 25: Comparison: Placebo vs CTP-543 8 mg BID; How Satisfied With Your Eyelashes: Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.3], Standard Error of Mean 0.10
Statistical Analysis 26: Comparison: Placebo vs CTP-543 12 mg BID; How Satisfied With Your Eyelashes: Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-0.8 to -0.4], Standard Error of Mean 0.11
Statistical Analysis 27: Comparison: Placebo vs CTP-543 8 mg BID; How Satisfied With Your Eyelashes: Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.5], Standard Error of Mean 0.11
Statistical Analysis 28: Comparison: Placebo vs CTP-543 12 mg BID; How Satisfied With Your Eyelashes: Week 16; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.7], Standard Error of Mean 0.12
Statistical Analysis 29: Comparison: Placebo vs CTP-543 8 mg BID; How Satisfied With Your Eyelashes: Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.5], Standard Error of Mean 0.11
Statistical Analysis 30: Comparison: Placebo vs CTP-543 12 mg BID; How Satisfied With Your Eyelashes: Week 20; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-1.0 to -0.5], Standard Error of Mean 0.12
Statistical Analysis 31: Comparison: Placebo vs CTP-543 8 mg BID; How Satisfied With Your Eyelashes: Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.6], Standard Error of Mean 0.12
Statistical Analysis 32: Comparison: Placebo vs CTP-543 12 mg BID; How Satisfied With Your Eyelashes: Week 24; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-1.2 to -0.7], Standard Error of Mean 0.13

15. Secondary Outcome: Change in the Anxiety and Depression Scale Scores of the Hospital Anxiety and Depression Scale (HADS) From Baseline at Week 24
Description: HADS is a questionnaire designed to assess anxiety and depression symptoms which is completed by participants. The questionnaire is comprised of two separate scales with a total of 14 items: A 7-item scale related to anxiety and 7-item scale related to depression. Each item within both scales is scored using a 4-point scale, ranging from 0 to 3 and the total scores in each scale can range from 0 to 21. Separate scores were created for anxiety and depression. A score between 0-7 is considered normal, 8-10 is mild, 11-14 is moderate, and >14 is severe anxiety or depression. Higher scores indicate greater severity. A negative change from baseline indicates less severity.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 128 | 318 | 200
score on a scale
  Anxiety: Baseline | 5.5 (3.92) | 6.2 (4.06) | 6.0 (3.92)
  Anxiety: Change From Baseline at Week 24 | -0.4 (2.98) | -1.0 (3.26) | -1.1 (3.24)
  Depression: Baseline | 3.3 (3.06) | 3.7 (3.31) | 3.6 (3.39)
  Depression: Change From Baseline at Week 24 | -0.7 (2.67) | -0.9 (2.93) | -1.1 (2.88)
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Anxiety; Test type: Superiority; p = 0.2489, ANCOVA — P-value was calculated by analysis of covariance (ANCOVA) analysis with effects for treatment, visit, baseline SALT score, and baseline HADS value; LS Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.9], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Anxiety; Test type: Superiority; p = 0.1235, ANCOVA — P-value was calculated by ANCOVA analysis with effects for treatment, visit, baseline SALT score, and baseline HADS value; LS Mean Difference = 0.5, 95% CI 2-sided [-0.1 to 1.1], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Placebo vs CTP-543 8 mg BID; Depression; Test type: Superiority; p = 0.9765, ANCOVA — [p-value comment as in outcome 15, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.25
Statistical Analysis 4: Comparison: Placebo vs CTP-543 12 mg BID; Depression; Test type: Superiority; p = 0.3559, ANCOVA — [p-value comment as in outcome 15, analysis 2]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.3 to 0.8], Standard Error of Mean 0.27

16. Secondary Outcome: Percentage of Participants Achieving an Absolute SALT Score of ≤10 at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 140 | 351 | 215
percentage of participants | 0 | 20.8 | 34.5
Statistical Analysis 1: Comparison: Placebo vs CTP-543 8 mg BID; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.21, 95% CI 2-sided [0.16 to 0.25], Standard Error of Mean 0.022
Statistical Analysis 2: Comparison: Placebo vs CTP-543 12 mg BID; Test type: Superiority; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 13, analysis 1]; Risk Difference (RD) = 0.33, 95% CI 2-sided [0.27 to 0.39], Standard Error of Mean 0.032

ADVERSE EVENTS:
Time Frame: All-cause mortality: Randomization up to Week 28; Adverse events: From first dose of study drug up to last follow up visit (Week 28)
Description: All-cause mortality: All randomized participants included all participants who were randomized in the study.
  Adverse events: Safety population included all participants who received study drug during the treatment period.
Arm/Group | Placebo | CTP-543 8 mg BID | CTP-543 12 mg BID
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/351 | 0/215
Serious Adverse Events (participants affected / at risk) | 4/140 | 4/350 | 1/215
Other Adverse Events (participants affected / at risk) | 31/140 | 117/350 | 75/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | CTP-543 8 mg BID (N=350) | CTP-543 12 mg BID (N=215)
Appendicitis (Infections and infestations) | 1 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | CTP-543 8 mg BID (N=350) | CTP-543 12 mg BID (N=215)
COVID-19 (Infections and infestations) | 8 | 19 | 15
Nasopharyngitis (Infections and infestations) | 5 | 18 | 8
Upper respiratory tract infection (Infections and infestations) | 9 | 9 | 8
Blood creatine phosphokinase (increased) (Investigations) | 2 | 21 | 11
Headache (Nervous system disorders) | 8 | 41 | 24
Acne (Skin and subcutaneous tissue disorders) | 7 | 31 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wants to publish study data or results, the publication or presentation must be provided to Concert for review at least 60 days in advance. If Concert needs to file a patent application prior to publication, the publication can be delayed up to 90 days from Sponsor providing notice to the investigator of such need.

DOCUMENTS (2):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT04518995/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT04518995/SAP_001.pdf